CLINICAL TRIAL: NCT03653585
Title: Cortical Lesions in the Primary Sensorimotor Hand Area and Their Impact on Dexterity in Multiple Sclerosis: a 7T MRI Study
Brief Title: Cortical Lesions in Patients With Multiple Sclerosis
Acronym: CLiMS
Status: Completed | Type: Observational
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: Scleroseforeningen (Unknown); Danish Multiple Sclerosis Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: CLiMS
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive
Keywords: Multiple Sclerosis; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Transcranial Magnetic Stimulation; Functional Neuroimaging; Cortical Lesion; Sensorimotor cortex; 7T; 7 Tesla
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lesion negative hemisphere in Healthy Controls (HC): Data grouped as an un-lesioned primary sensorimotor cortical hemisphere in age and sex matched healthy voluntary participants
- Lesion negative hemisphere in patients (PT-N): Data grouped as an un-lesioned primary sensorimotor cortical hemisphere in MS patients
- Lesion positive hemisphere in patients (PT-P): Lesion positive hemisphere in patients:
  Data grouped as a lesioned primary sensorimotor cortical hemisphere in MS patients

SUMMARY:
Multiple sclerosis (MS) is an autoimmune disease, leading to inflammation and degeneration of neurons in the entire central nervous system (CNS). Not only does MS attack CNS white matter, the wiring of the brain, but it also affects so called grey matter, involved in communication between brain cells. Some studies have shown that grey matter damage and lesions to the outermost layer of the brain, the cortex, might serve as a better diagnostic and prognostic tool for MS patients. The issue is that cortical lesions only to a limited extent can be visualized by conventional magnetic resonance imaging (MRI) at 3 tesla. The new generation of ultra-high field MR scanners with a field strength of 7 tesla, has a higher sensitivity towards detecting these cortical lesions. We therefore wish to use the improved sensitivity of ultra-high field MRI to improve detection of cortical lesions, and to elucidate the detrimental effects of single lesions to the cortex, thereby improving both diagnosis and prognosis of the disease.

By implementing newly developed ultra-high-resolution MR-sequences the amount and extent of cortical lesions to the area of the brain responsible of the sensory and motor function of the hand (sensorimotor hand area - SM1-HAND) will be investigated in patients with relapsing remitting and secondary progressive MS. We will also assess how these lesions affect manual dexterity and sensory function and how cortical lesions affect communication within brain areas. It is hypothesized that the amount and size of cortical lesions is highly involved in brain communication and manual function, a major problem in MS, and that this project will shed new light on how the disease damages this important brain area.

DETAILED DESCRIPTION:
BACKGROUND. In recent years, several lines of research have shown that multiple sclerosis (MS) affects cortical grey matter and that the degree of cortical grey matter involvement is associated with cognitive and physical disability, but the specific impact of a cortical lesion on regional function remains to be clarified.

High-field Magnetic Resonance Imaging (MRI) at 3T has been used to detect cortical lesions in MS, but histological examinations have shown that only 'the tip of the iceberg' is detected. Ultra-high field 7T MRI has a higher diagnostic sensitivity than 3T MRI. Although not every cortical lesion is detected even at 7T, a recent post-mortem verification study concluded that ultra-high field MRI "more than doubles detection of cortical MS lesions, compared to 3T MRI". Implementing 7T MRI in detection of cortical lesions and elucidating the behavioural and neurophysiological impact of cortical lesions is therefore a good candidate in aiding to resolve the clinico-radiological paradox reported in MS.

AIMS and HYPOTHESES. This study is designed to clarify the occurence of cortical lesions within the primary sensory-motor hand area (SM1-HAND) and their impact on manual motor and sensory function, as well as regional cortical connectivity. The SM1-HAND is well suited to address this question, because functional integration in SM1-HAND can be studied in detail with transcranial magnetic stimulation (TMS) and high-resolution fMRI.

Exploiting the increased sensitivity of 7T MRI to detect cortical lesions, the number, size and regional distribution of cortical lesions in SM1-HAND will be assessed and lesion load in SM1-HAND will be related to MRI-based, electrophysiological, and behavioral correlates of hand function.

Specifically the following parameters will be assessed:

1. The extent that the primary sensorimotor cortex is affected by cortical lesions in patients with relapsing remitting and secondary progressive multiple sclerosis (MS).
2. The impact of a single cortical MS lesion in the sensorimotor cortex on upper extremity sensorimotor function.
3. The impact of a single cortical MS lesion in the sensorimotor cortex on regional intra-cortical connectivity.

Hypotheses:

1) The extent of cortical damage to the primary sensorimotor cortex is unknown, but based on clinical symptoms of motor function it is expected that up to 40% of patients show focal cortical lesions in this area and that this will include all subtypes of cortical lesions.

2a) It is hypothesized that unimanual motor function correlates negatively with the total cortical lesion load within the contralateral sensorimotor cortex, independent of age, gender, handedness, white matter lesion volume, axonal integrity of the cortico-spinal tract, central motor conduction time and cortical thickness of the sensorimotor cortex. 2b) It is hypothesized that the amount and size of cortical lesions within the primary sensorimotor cortex correlates positively with motor fatigue. 2c) It is hypothesized that unimanual sensory acuity correlates negatively with the total cortical lesion load within the contralateral sensorimotor cortex.

3a) It is expected cortical lesions to cause a shift in the digit representation, measured as the task related BOLD signal of the contralateral somatosensory cortex, away from the lesion. 3b) It is hypothesized that cortical lesions within the primary sensorimotor cortex affects the regional intra-cortical excitatory/inhibitory balance.

4) It is further expected that the functional impact of regional cortical lesions are independent of age, gender, handedness, white matter lesion volume, axonal integrity of the cortico-spinal tract, central motor conduction time and cortical thickness of the sensorimotor cortex and scales with lesion type, number and volume.

3. RESEARCH PLAN.

Part 1. Whole-brain 7T MRI study to identify cortical lesions.

Participants: The project is planned to involve 80 mildly to moderately affected patients (Expanded Disability Status Scale of <5.5) with relapsing-remitting MS (RR-MS, n=40) or secondary progressive MS (SP-MS, n=40) who had no clinical relapse within the last three months and 20 healthy age-matched controls (age range: 18-70 years).

Ultra-high field MRI. All participants will be studied with whole-brain ultra-high field MRI at 7T, using a research-only 7T Achieva MR system (Philips, Best, The Netherlands) located at Hvidovre Hospital. Whole-brain MR scanning will be performed with a dual transmit, 32-channel receive head coil (Nova Medical Products), including 3-dimensional (3-D), magnetization-prepared rapid acquisition of gradient echoes (MPRAGE) imaging at 0.65-mm isotropic resolution and 3-D, magnetization-prepared, fluid attenuated inversion recovery (MPFLAIR) imaging at 0.7-mm isotropic resolution (5). Whole-brain semi-quantitative (MP2RAGE), as well as a quantitative T2* sequence will also be conducted.

Additional examinations. Outside the MR scanner, physical impairment (EDSS), fatigue (Fatigue Scale for Motor and Cognitive Functions, FSMC), cognition (Symbol Digit Modalities Test, SMDT & Paced Auditory Serial Addition Test, PASAT), depression (Beck Depression Inventory, BDI II) as well as sensorimotor hand function (9HPT, Jebsen Taylor Hand Function Test (JTT), Finger tapping, Grating Orientation Discrimination Test (GODT)) will be assessed.

Part 2. Selected 7T MRI of the SM1-HAND.

Participants: A sub-group of individuals who participated in part 1 will be asked to participate in part 2: It is expected that at least 20 patients will show at least one cortical lesion in the right or left SM1-HAND on 7T MRI. The lesion-positive patients (n>20), an age- and EDSS- matched lesion-negative MS group (n>20), and an age-matched healthy control group (n=20) will be studied. Recruitment will be done continuously to minimize the delay between part 1 & 2.

Participants will be scanned again with the 7T Achieva MR system using a reduced coronal field-of-view, covering the right and left SM1-HAND and the corticospinal tract. Structural imaging will include a 0.7 mm isotropic FLAIR sequence, and an ultra-high resolution MP2RAGE (0.5 mm isotropic) sequence as well as whole brain diffusion weighted imaging (DWI). Proton-Magnetic Resonance Spectroscopy (MRS) will be performed to measure regional N-acetyl-aspartate (NAA), GABA and glutamate concentration in right and left SM1-HAND. Lastly high-spatial resolution functional Blood Oxygen Level Dependent (BOLD) (fMRI) will be used to map the somatotopy of sensory and motor representations in SM1-HAND. Activation maps will be superimposed to individual lesion maps.

TMS. The corticospinal conduction will be quantified with transcranial magnetic stimulation (TMS). A novel neuronavigated TMS mapping method developed by this group, which is sensitive to changes in cortico-motor representations of intrinsic hand muscles will also be implemented. Finally, aspects of intracortical inhibition in both SM1-HAND with established single-pulse and double-pulse TMS paradigms will be carried out. Conduction in the afferent somatosensory pathway will be assessed by recording somatosensory evoked potentials (SSEP).

ELIGIBILITY:
Inclusion Criteria:

Patients

* Expanded Disability Status Scale of < 7.5
* Diagnosed with either relapsing-remitting or secondary progressive multiple sclerosis
* No clinical relapse within last three months
* Have the ability to comply with all requirements of the study protocol, as determined by the investigator

Healthy controls

* Able bodied
* Have the ability to comply with all requirements of the study protocol, as determined by the investigator

Exclusion Criteria:

Patients

* Pregnancy
* Pacemaker or other implanted electronic devices
* Claustrophobia
* Psychiatric disorder
* Administration of acute cortisol
* Changes in pharmacological treatment within the last 3 months
* Close relatives suffering from epilepsy (only relevant for TMS)
* Migraine (only relevant for TMS)
* Any contraindication to TMS or MRI
* Persons who do not wish to be informed about abnormal findings as part of the investigations

Healthy controls

* Pregnancy
* Under medication at the time of the experiment (with the exception of contraceptive drugs)
* History of neurologic disease
* Pacemaker or other implanted electronic devices
* Close relatives suffering from epilepsy (only relevant for TMS)
* Migraine (only relevant for TMS)
* History of cerebral hemorrhage or brain damage
* Claustrophobia
* Psychiatric disorder
* Any contraindication to TMS or MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 40 healthy control volunteers will be recruited from the general population via the departments webpage (www.drcmr.dk), publicly available advertising media 'http://www.forsoegsperson.dk/', links on social media portal: 'facebook' and advertisements in newsstands and communication-boards in public facilities like canteens, educational institutions, sports facilities and hospitals in the Copenhagen area.
  Recruitment of 80 patients will in addition be done through the ambulatory care at the Danish Multiple Sclerosis Centre (DMSC) at Rigshospitalet in Copenhagen, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Number of cortical lesions in the primary sensorimotor cortex (SM1) | Data collected on day 1 and 2
  Quantified as cortical lesion number on a unihemispheric level in patients with relapsing remitting and secondary progressive multiple sclerosis (RRMS & SPMS)
  The extent of damage to the SM1 is unknown, but based on clinical symptoms of motor function we expect that up to 40% of patients show focal cortical lesions in this area.
  Additionally we wish to explore the relationship between cortical lesions in SM1 and other MRI metrics (e.g. white matter lesion load of the cortico-spinal tract, cortical myelination, cortical thickness, metabolite levels of SM1-HAND and diffusion metrics of the cortico-spinal tract)
Unimanual motor function | Data acquired on day 1
  A composite score computed as the mean of Z-scores from the health population (expected range +-4, lower being better motor performance) for unimanual performance in: 9-hole peg test (time in seconds, lower being better), Jebsen Taylor Hand Function Test (time in seconds, lower being better), Finger Tapping (mean times/10seconds from all 5 digits, higher being better).
  We hypothesize that unimanual motor function correlates negatively with the total cortical lesion load within the contralateral SM1-HAND area, independent of age, gender handedness, white matter lesion volume and axonal integrity of the cortico-spinal tract, central motor conduction time (CMCT) and cortical thickness of the primary sensorimotor cortex.

SECONDARY OUTCOMES:
Functional brain activation pattern as revealed by task related blood oxygenation level dependent (BOLD) signal changes. | Data acquired on day 2
  Measured as the digit specific BOLD signal from the contralateral SM1 during vibrotactile digit stimulation and 1 Hz finger tapping of each digit.
  We expect that the presence of at cortical lesion will cause a spatial shift in digit representation away from the lesion, affect the area of activation and overlap of activation patterns between digits.
Unimanual sensory acuity | Data acquired on day 1
  Quantified as a composite score computed as mean of Z-scores across the entire population (expected range +-4, higer being better) derived from the unimanual performance in the grating orientation discrimination task (GODT, discrimination distance in mm, range 0.5 to > 3, lower being better) and the sum of functional systems sensory score from each individual digit (range 0-6, lower being better)
  We expect unimanual sensory acuity to be correlated negatively with cortical lesion volume of the primary sensory cortex and digit specific BOLD signal derived from the fMRI BOLD activation map from vibrotactile stimulation.
Intra-cortical inhibition and facilitation (Exploratory outcome measure) | Data acquisition on day 3
  Measured, using transcranial magnetic stimulation (TMS), as short interval intra-cortical inhibition (SICI) and intra-cortical facilitation (ICF), short afferent inhibition (SAI) and short afferent facilitation (SAF), cortical silent period (CSP) and Ipsilateral silent period (iSP).
  And as regional GABA and glutamate concentrations, using magnetic resonance spectroscopy (MRS).
  We hypothesize that cortical lesions in the SM1 will alter the regional intra-cortical inhibitory/excitatory balance evident as changes in TMS derived measures of intra-cortical inhibition and facilitation and that this correlates with regional changes in GABA and Glutamate measured with MRS.
Regional NAA concentration of the SM1 | Data acquired on day 2
  Measured as NAA concentration derived from MRS of a 2x2x2 voxel of the primary sensorimotor hand area.
  We expect NAA concentration within a lesioned hemisphere to be decreased and to correlate with unimanual motor function and sensory acuity.
Cortical lesion subtype (Exploratory outcome measure) | Data acquisition on day 1 and 2
  Cortical lesions within in the SM1 will be qualitatively determined, using conventional standards, as either juxtacortical, leukocortical, intracortical or subpial.
  We wish to explore how lesion subtype influences our primary and secondary outcome measures.
Expanded Disability status scale (EDSS) score | Data collected on day 1
  EDSS (range 0-10, lower being better) score determined by neurological examination
  We expect EDSS score to be correlated positively with whole brain cortical lesion volume independent of our covariates
Motor fatigue | Assessed on day 1
  Motor fatigue score (range 10-50, lower being better) from the Fatigue Scale for Motor and Cognitive Functions (FSMC) questionnaire.
  We hypothesize that the amount and size of cortical lesions within the primary sensorimotor cortex correlates positively with motor fatigue.
Volume of cortical lesions in the primary sensorimotor cortex (SM1) | Data collected on day 1 and 2
  Quantified as the volume for cortical lesions within the cortex on a unihemispheric level in patients with RRMS or SPMS.
  We hypothesize that the volume of cortical lesions has a negative impact on sensory and motor function of the contralateral hand

OTHER OUTCOMES:
MRI metrics (Exploratory outcome measure) | Data is collected at a single time point during either the first, second and third day of the experiment
  Unrelated to the primary hypotheses of this study, the collected MRI metrics allow for further exploratory analysis for future hypothesis formulation.
  This involves e.g. investigation of a relationship between white matter damage and cortical lesions. Exploration the relationship between cortical lesions and subpial demyelination. The presence of central veins within cortical lesion subtypes.
Cognition | Assessed on day 1
  Composite score of computed as the mean of Z-scores (expected range +-4, higher being better) from the population for the paced auditory serial addition test (PASAT, number of correct answers, range 0-60, higher being better) and symbol digit modalities test (SDMT, number of correct responses, range 0-110, higher being better)
Depression | Assessed on day 1
  Depression score from the Beck depression inventory II (BDI-II) questionnaire (range 0-63, lower being less depressed).
Cortical thickness of the primary sensorimotor cortex. (Covariate) | Acquired on day 1
  Cortical thickness of the SM1 measured in mm from segmented MR images
White matter lesion load of the corticospinal tract. (Covariate) | Acquired on day 1
  Total volume of white matter lesions in the corticospinal tract
Handedness (covariate) | Acquired on day 1
  Laterality index (range +-100, higher being more right handed) derived from the Oldfield handedness inventory questionnaire.
Corticomotor conduction time (CMCT) (covariate) | Acquired on day 3
  Quantified as time (in ms)
White matter integrity of the corpus callosum and the corticospinal tract (Covariate) | Acquired on day 2
  Measured using established diffusion tensor imaging metrics.
Total white matter lesion load (covariate) | Acquired on day 1
  Whole brain volume of white matter lesions
Whole brain cortical volume (covariate) | Acquired on day 1
  Volume of cortical greymatter derived from segmented MR images

CONTACTS AND LOCATIONS:
Overall Officials: Hartwig R Siebner, Professor, Principal Investigator — Danish Research Centre for Magnetic Resonance
Locations (1):
- Danish Research Centre for Magnetic Resonance, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to Danish data protection legislation, it is currently not allowed to publish individual participant data.
  Data that underlie published results related to the primary and secondary outcome measures will, following anonymization, be made publicly available. However, data will be grouped in appropriate age categories with minimum 5 participants in each group.

REFERENCES:
- [Background] Harrison DM, Roy S, Oh J, Izbudak I, Pham D, Courtney S, Caffo B, Jones CK, van Zijl P, Calabresi PA. Association of Cortical Lesion Burden on 7-T Magnetic Resonance Imaging With Cognition and Disability in Multiple Sclerosis. JAMA Neurol. 2015 Sep;72(9):1004-12. doi: 10.1001/jamaneurol.2015.1241. PMID 26192316
- [Background] Nielsen AS, Kinkel RP, Madigan N, Tinelli E, Benner T, Mainero C. Contribution of cortical lesion subtypes at 7T MRI to physical and cognitive performance in MS. Neurology. 2013 Aug 13;81(7):641-9. doi: 10.1212/WNL.0b013e3182a08ce8. Epub 2013 Jul 17. PMID 23864311
- [Background] Calabrese M, Poretto V, Favaretto A, Alessio S, Bernardi V, Romualdi C, Rinaldi F, Perini P, Gallo P. Cortical lesion load associates with progression of disability in multiple sclerosis. Brain. 2012 Oct;135(Pt 10):2952-61. doi: 10.1093/brain/aws246. PMID 23065788
- [Background] de Graaf WL, Kilsdonk ID, Lopez-Soriano A, Zwanenburg JJ, Visser F, Polman CH, Castelijns JA, Geurts JJ, Pouwels PJ, Luijten PR, Barkhof F, Wattjes MP. Clinical application of multi-contrast 7-T MR imaging in multiple sclerosis: increased lesion detection compared to 3 T confined to grey matter. Eur Radiol. 2013 Feb;23(2):528-40. doi: 10.1007/s00330-012-2619-7. Epub 2012 Aug 17. PMID 22898935
- [Background] Kilsdonk ID, Jonkman LE, Klaver R, van Veluw SJ, Zwanenburg JJ, Kuijer JP, Pouwels PJ, Twisk JW, Wattjes MP, Luijten PR, Barkhof F, Geurts JJ. Increased cortical grey matter lesion detection in multiple sclerosis with 7 T MRI: a post-mortem verification study. Brain. 2016 May;139(Pt 5):1472-81. doi: 10.1093/brain/aww037. Epub 2016 Mar 8. PMID 26956422
- [Background] Raffin E, Pellegrino G, Di Lazzaro V, Thielscher A, Siebner HR. Bringing transcranial mapping into shape: Sulcus-aligned mapping captures motor somatotopy in human primary motor hand area. Neuroimage. 2015 Oct 15;120:164-75. doi: 10.1016/j.neuroimage.2015.07.024. Epub 2015 Jul 15. PMID 26188259
- [Background] Kujirai T, Caramia MD, Rothwell JC, Day BL, Thompson PD, Ferbert A, Wroe S, Asselman P, Marsden CD. Corticocortical inhibition in human motor cortex. J Physiol. 1993 Nov;471:501-19. doi: 10.1113/jphysiol.1993.sp019912. PMID 8120818
- [Background] Dubbioso R, Raffin E, Karabanov A, Thielscher A, Siebner HR. Centre-surround organization of fast sensorimotor integration in human motor hand area. Neuroimage. 2017 Sep;158:37-47. doi: 10.1016/j.neuroimage.2017.06.063. Epub 2017 Jun 29. PMID 28669907